CLINICAL TRIAL: NCT01151319
Title: A Randomized Single-blind Placebo-controlled Study to Evaluate the Safety and Immunogenicity of Three Candidate HIV-1 Vaccines, pSG2.HIVconsv DNA, ChAdV63.HIVconsv and MVA.HIVconsv, Administered in Combination to Healthy HIV 1 Uninfected Adults
Brief Title: Safety and Immunogenicity Study of Three Candidate HIV-1 Vaccines, Administered in Combination to Healthy HIV-1 Uninfected Adults
Acronym: HIV-CORE 002
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HIV-CORE 002
Record Dates: First submitted 2010-06-24; First posted 2010-06-28 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-04

CONDITIONS: HIV-1 Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Stage 1. (Experimental): The first stage will start from a low and well tolerated, but likely less immunogenic dose of ChAdV63.HIVconsv (n=2).
  Interventions: Biological: ChAdV63.HIVconsv low dose.
- Stage 2 (Experimental): The highest dose of ChAdV63.HIVconsv followed by boost with MVA.HIVconsv at week 0 and 8, respectively (n=8). Followed up at 6,12 and 24 months after last vaccination.
  Interventions: Biological: ChAdV63.HIVconsv high dose.; Biological: MVA.HIVconsv
- Stage 3 (Experimental): Three doses of pSG2.HIVconsv DNA followed by boost with high dose ChAdV63.HIVconsv followed by boost with MVA.HIVconsv at week 0,4,8,12 and 20, respectively (n=8). Followed up at 6, 12 and 24 months after last vaccination.
  Interventions: Biological: ChAdV63.HIVconsv high dose.; Biological: pSG2.HIVconsv; Biological: MVA.HIVconsv
- Stage 4 (Experimental): Three doses of pSG2.HIVconsv DNA followed by boost with MVA.HIVconsv followed by boost with high dose ChAdV63.HIVconsv at weeks at week 0,4,8,12 and 16, respectively (n=8).
  Interventions: Biological: ChAdV63.HIVconsv high dose.; Biological: pSG2.HIVconsv; Biological: MVA.HIVconsv
- Stage 2 Placebo (Placebo Comparator): Time-course matched to vaccinations (n=2)
  Interventions: Other: Placebo
- Stage 3 placebo (Placebo Comparator): Time-course matched to vaccinations (n=2)
  Interventions: Other: Placebo
- Stage 4 placebo (Placebo Comparator): Time-course matched to vaccinations (n=2)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: ChAdV63.HIVconsv low dose. — Attenuated chimp adenovirus. 5x10^9 virus particles.
  Arms: Stage 1.
Biological: ChAdV63.HIVconsv high dose. — Attenuated chimp adenovirus at 5x10^10 virus particles.
  Arms: Stage 2; Stage 3; Stage 4
Biological: pSG2.HIVconsv — DNA at 4mg per dose.
  Arms: Stage 3; Stage 4
Biological: MVA.HIVconsv — Attenuated poxvirus at 4x10^8 plaque forming units per dose.
  Arms: Stage 2; Stage 3; Stage 4
Other: Placebo — Phosphate buffered saline
  Arms: Stage 2 Placebo; Stage 3 placebo; Stage 4 placebo

SUMMARY:
This is a randomised, placebo-controlled, single-blind study designed to evaluate the safety and immunogenicity of three novel HIV vaccines.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or females, as assessed by a medical history, physical examination and laboratory tests.
2. Aged at least 18 years on the day of screening and no greater than 50 years on the day of the first vaccination.
3. Willing to comply with the requirements of the protocol and available for follow-up for the planned duration of the study.
4. In the opinion of the principal investigator or designee, the volunteer has understood the information provided. Written informed consent must be given before any study-related procedures are performed.
5. Willing to undergo HIV-1 testing, HIV-1 counselling and receive HIV-1 test results.
6. If heterosexually active female; using an effective method of contraception (e.g. hormonal contraception, diaphragm, intra-uterine device (IUD), condoms, anatomical sterility in self or partner) from 14 days prior to the first vaccination until at least 6 weeks after the last vaccination; all female volunteers must be willing to undergo urine pregnancy tests at time points specified in the protocol.
7. If heterosexually active male; willing to use an effective method of contraception (condoms; anatomical sterility in self or partner) from the day of the first vaccination until 6 weeks after the last vaccination.
8. Willing to forgo donations of blood during the study.

Exclusion Criteria:

1. Any clinically significant acute or chronic medical condition that is considered progressive or, in the opinion of the principal investigator or designee, would make the volunteer unsuitable for the study.
2. Any of the following abnormal laboratory parameters listed below:

   Haematology
   * Haemoglobin < 10.0 g/dl
   * Absolute Neutrophil Count (ANC) ≤ 1000 /mm3 (≤ 1 x 109 /l)
   * Absolute Lymphocyte Count (ALC) ≤ 600 /mm3 (≤ 1 x 109 /l)
   * Platelets ≤100,000 /mm3, ≥ 550,000 /mm3 (≤ 90 /l, ≥ 550 /l) Biochemistry
   * Creatinine > 1.3 x ULN
   * Aspartate aminotransferase (AST) > 2.5 x ULN
   * Alanine aminotransferase (ALT) > 2.5 x ULN Urinalysis
   * Abnormal dipstick confirmed by microscopy
3. Reported high-risk behaviour for HIV infection. High-risk behaviour for HIV-1 infection is defined as follows. Within the previous 6 months the volunteer has:

   * Had unprotected vaginal or anal sex with a known HIV-infected person or a casual partner (i.e., no continuing, established relationship)
   * Engaged in sex work for money or drugs
   * Used injection drugs
   * Acquired one of the following sexually transmitted disease (STD); Chlamydia, gonorrhoea and syphilis.
4. Confirmed HIV-1 or HIV-2 infection.
5. If female, pregnant or planning a pregnancy within 6 weeks after last vaccination; or lactating.
6. Receipt of live attenuated vaccine within the previous 60 days (live attenuated flu vaccine within 14 days) or planned receipt within 60 days after vaccination with Investigational Product or receipt of other vaccine within the previous 14 days or planned receipt within14 days after vaccination with Investigational Product.
7. Receipt of blood transfusion or blood products within the previous 6 months.
8. Participation in another clinical trial of an Investigational Product currently, within the previous 3 months or expected participation during this study.
9. Receipt of any investigational HIV vaccine within the last 6 years.
10. History of severe or very severe local or systemic reactogenicity events, or history of severe or very severe allergic reactions.
11. Confirmed diagnosis of hepatitis B virus (surface antigen, HBsAg), hepatitis C virus (HCV antibodies) or active syphilis.
12. Smallpox vaccination within the previous 3 years (smallpox vaccination prior to 3 years should be documented but is not an exclusion criterion).
13. Major psychiatric illness including any history of schizophrenia or severe psychosis, bipolar disorder requiring therapy, suicidal attempt or ideation in the previous 3 years.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2010-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Safety | Actively collected data throughout the study until 6 months after the last vaccination
  Proportion of volunteers who develop a grade 3 or 4 local reaction.

SECONDARY OUTCOMES:
Immunogenicity | Samples will be collected at every visit pre- and post vaccination
  Proportion of volunteers who develop new CD8+ and CD4+ T cell responses to one or more HIV-1 epitopes, as determined by IFN-γ ELISPOT assay.
Immunogenicity | Stage 1; screen, 0, 1, 2, 4, 8, 16, 28 wk. Stage 2; screen, 0, 1, 2, 4, 8, 9, 12, 20, 28 wk. Stage 3; screen, 1, 8, 12, 13, 14, 20, 21, 22, 28 wk. Stage 4; screen, 0, 8, 12, 13, 16, 17, 18, 24, 28 wk post vac. Stage 2 & 3: 6,12,24 mth after last vaccine
  Exploration of the efficacy of vaccine-induced CD8+ T cells to suppress HIV-1 replication in vitro.

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Hanke, Principal Investigator — University of Oxford; Lucy Dorrell, Principal Investigator — University of Oxford
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine, Oxford, Oxon, United Kingdom

REFERENCES:
- [Derived] Moyo N, Borthwick NJ, Wee EG, Capucci S, Crook A, Dorrell L, Hanke T. Long-term follow up of human T-cell responses to conserved HIV-1 regions elicited by DNA/simian adenovirus/MVA vaccine regimens. PLoS One. 2017 Jul 18;12(7):e0181382. doi: 10.1371/journal.pone.0181382. eCollection 2017. PMID 28719652
- [Derived] Borthwick N, Lin Z, Akahoshi T, Llano A, Silva-Arrieta S, Ahmed T, Dorrell L, Brander C, Murakoshi H, Takiguchi M, Hanke T. Novel, in-natural-infection subdominant HIV-1 CD8+ T-cell epitopes revealed in human recipients of conserved-region T-cell vaccines. PLoS One. 2017 Apr 27;12(4):e0176418. doi: 10.1371/journal.pone.0176418. eCollection 2017. PMID 28448594
- [Derived] Hayton EJ, Rose A, Ibrahimsa U, Del Sorbo M, Capone S, Crook A, Black AP, Dorrell L, Hanke T. Safety and tolerability of conserved region vaccines vectored by plasmid DNA, simian adenovirus and modified vaccinia virus ankara administered to human immunodeficiency virus type 1-uninfected adults in a randomized, single-blind phase I trial. PLoS One. 2014 Jul 9;9(7):e101591. doi: 10.1371/journal.pone.0101591. eCollection 2014. PMID 25007091